CLINICAL TRIAL: NCT05960123
Title: Evaluation of TIP Urethroplasty With Spongioplasty-Dartosoraphy Reinforcement in Pediatric Hypospadias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohammad Daboos, Professor of pediatric surgery, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 0000395-24-01-019
Record Dates: First submitted 2023-07-10; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Hypospadias; Complication,Postoperative
Keywords: Distal and midpenile hypospadias; TIPU; Spongioplasty-dartosoraphy; pediatric HOSE
MeSH Terms: conditions — Hypospadias; Postoperative Complications | interventions — Lysine Acetyltransferase 5

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with Spongioplasty (Active Comparator): patients underwent TIPU with spongioplasty-Dartosoraphy reinforcement
  Interventions: Procedure: Tubularized Incised Plate (TIP) urethroplasty
- Group without Spongioplasty (Active Comparator): patients underwent TIPU with dorsal dartos flap interposition without spongioplasty
  Interventions: Procedure: Tubularized Incised Plate (TIP) urethroplasty

INTERVENTIONS:
Procedure: Tubularized Incised Plate (TIP) urethroplasty — tubularization of urethral plate with or without spongioplasty

SUMMARY:
The study aimed to evaluation of Tubularized incised palate urethroplasty with spongioplasty-dartosoraphy reinforcement (group A) through comparing of functional and cosmetic results of this technique with the conventional TIP urethroplasty (group B).

ELIGIBILITY:
Inclusion Criteria:

* lees than 14 years Distal hypospadias urethral plate size more than 6mm glans size more than 14 mm

Exclusion Criteria:

* recurrent cases Proximal; hypospadias

Ages: 6 Months to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — this anomalies of male genitalia
Enrollment: 220 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Urethrocutaneous fistula | 12 months
  Rate of fistula
meatal stenosis | 12 months
  Rate of metal stenosis
glans dehiscence | 12 months
  Rate of glans dehiscence

OTHER OUTCOMES:
Cosmetic results | 12 months
  Hypospadias Objective Scoring Evaluation (maximum the best is 16 points ) and minimum the worst is 4

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Daboos, Cairo, Select, Egypt

IPD SHARING:
Plan to Share IPD: No